CLINICAL TRIAL: NCT06336993
Title: Traditional Chinese Herbal Compound as Complementary Treatment for Non-specific Low Back Pain: A Randomized Controlled Trail Study
Brief Title: Evaluation of Clinical Efficacy of Herbal Compound in the Treatment of NSLBP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Principal Investigator, Yangjun Lao, Zhejiang Traditional Chinese Medicine Science and Technology Plan Project Leader, Zhejiang Provincial Tongde Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: liuxianguiji
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- herbal compound (Experimental)
  Interventions: Drug: herbal compound
- celecoxib (Active Comparator)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: herbal compound — patients were instructed to take the herbal compound twice a day for 3 weeks, 200 to 300ml each time, composition of herbal compound of BSTL was BaiShao 9g, ChuanNiuXi 15g, DanShen 15g, DiLong 9g, DuHuo 9g, DuZhong 15g, GouJi 15g, QinJiao 9g, SangJiSheng 15g, XiXianCao 9g, XuChangQin 9g and YanHuSuo 9g, and herbs were provided by the Traditional Chinese Medicine pharmacy of Tongde Hospital in Zhejiang Province.
  Arms: herbal compound
Drug: Celecoxib — Celecoxib (Ouyi Pharmaceutical Co., LTD., H20203296) was used twice a day for 3 weeks, 200mg/ time, to treat NSLBP;
  Arms: celecoxib

SUMMARY:
The aim of this randomized controlled trial was to explore the clinical efficacy and safety of HXTL in the treatment of NSLBP based on TCM principles and to compare the clinical outcomes of different syndromes of NSLBP with celecoxib.In this study, 80 patients with NSLBP were recruited and randomly grouped to use TCM compound and celeoxib respectively for intervention. The pain status and lumbar function use scale of patients were scored before intervention, 1 week, 2 weeks and 3 weeks after intervention, and the adverse reactions of patients after medication were recorded, and the clinical efficacy of the two groups of patients was compared finally.

ELIGIBILITY:
Inclusion Criteria:

* a. Patients with low back pain who were seen between January 1, 2022 and June 16, 2023 were included;
* b. meet the diagnostic criteria of NSLBP;
* c. the age range was 20-90 years old;
* d. agree to participate in the study and sign the informed consent;

Exclusion Criteria:

* a. those who are unable to communicate normally, such as those suffering from mental and cognitive diseases, and cannot cooperate with the treatment;
* b. pregnant or lactating women;
* c. patients who are allergic to the treatment components or sulfonamides;
* d. patients with a history of coronary artery bypass grafting;
* e. patients with active gastrointestinal ulcer or bleeding;
* f. patients with severe heart failure;
* g. Patients with hepatic and renal insufficiency.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | baseline, 1 week, 2 week, 3 week after treating
  The visual analogue scale (VAS) is used to assess pain. It is widely used in clinical practice worldwild. The basic method is to use a walking scale about 10cm long, marked with 10 scales on one side, and the two ends are respectively "0" and "10". 0 indicates no pain, and 10 indicates the most unbearable pain. A higher score means more intense pain.
Oswestry disability index | baseline, 1 week, 2 week, 3 week after treating
  The Oswestry Disability Index (ODI) consists of 10 questions about pain intensity, self-care, lifting, walking, sitting, standing, disturbance of sleep, sexual life, social life, and travel, with six options for each question. The maximum score for each question is 5. Select the first option to score 0 points, select the last option to score 5 points, if there are 10 questions have been answered, the scoring method is: actual score /50 (highest possible score) × 100%, if there is a question not answered, the scoring method is: Actual score /45 (highest possible score) x 100%, if higher indicates more severe dysfunction.
Japanese Orthopaedic Association Scores | baseline, 1 week, 2 week, 3 week after treating
  Japanese Orthopaedic Association Scores are evaluated from four aspects: conscious symptoms, objective examination, limit of daily activities and bladder function. Each part is composed of several questions, with 3-4 options for each question. The highest score for each question is 2 or 3 points. The overall score ranges from 0 to 29, with lower scores indicating greater dysfunction.

OTHER OUTCOMES:
the adverse reactions of digestive or other system | baseline, 1 week, 2 week, 3 week after treating
  If the patient has a digestive or systemic adverse reaction, the patient's specific symptoms and timing will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Tongde Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Result] Bernstein IA, Malik Q, Carville S, Ward S. Low back pain and sciatica: summary of NICE guidance. BMJ. 2017 Jan 6;356:i6748. doi: 10.1136/bmj.i6748. No abstract available. PMID 28062522
- [Result] Oltean H, Robbins C, van Tulder MW, Berman BM, Bombardier C, Gagnier JJ. Herbal medicine for low-back pain. Cochrane Database Syst Rev. 2014 Dec 23;2014(12):CD004504. doi: 10.1002/14651858.CD004504.pub4. PMID 25536022
- [Result] Zhan JW, Li KM, Zhu LG, Wang SQ, Feng MS, Wei X, Yu J, Tang B, Yin XL, Han T, Zhang P, Li LH, Chen M, Shao CC. Efficacy and Safety of Bushen Huoxue Formula in Patients with Discogenic Low-Back Pain: A Double-Blind, Randomized, Placebo-Controlled Trial. Chin J Integr Med. 2022 Nov;28(11):963-970. doi: 10.1007/s11655-022-3505-4. Epub 2022 Jul 15. PMID 35840851